CLINICAL TRIAL: NCT03131648
Title: A Randomised, Double-blind, Placebo-controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Tralokinumab Monotherapy in Subjects With Moderate to Severe Atopic Dermatitis Who Are Candidates for Systemic Therapy
Brief Title: Tralokinumab Monotherapy for Moderate to Severe Atopic Dermatitis - ECZTRA 1 (ECZema TRAlokinumab Trial no. 1)
Acronym: ECZTRA 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1325; 2016-004200-65 (EudraCT Number)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor any of the investigator or LEO staff who are involved in the treatment or clinical evaluation and monitoring of the subjects will be aware of the treatment received. The packaging and labelling of the IMPs will contain no evidence of their identity.
  Since tralokinumab and placebo are visually distinct and not matched for viscosity, IMP will be handled and administered by a qualified, unblinded HCP at the site who will not be involved in the management of trial subjects and who will not perform any of the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Initial treatment period - Tralokinumab Q2W (Experimental): Week 0 to Week 16:
  Two subcutaneous (SC) injections of tralokinumab as a loading dose on Day 0, followed by a SC injection of tralokinumab Q2W regimen for 16 weeks.
  Interventions: Drug: Tralokinumab
- Initial treatment period - Placebo Q2W (Placebo Comparator): Week 0 to Week 16:
  Two subcutaneous (SC) injections of placebo as a loading dose on Day 0 followed by a SC injection of placebo Q2W regimen for 16 weeks.
  Interventions: Drug: Placebo
- Maintenance treatment period - Tralokinumab Q2W (Experimental): Week 16 to Week 52:
  Tralokinumab responders from the initial treatment period re-randomised at Week 16 and administered tralokinumab maintenance subcutaneous injection regimen Q2W for 36 weeks.
  Interventions: Drug: Tralokinumab
- Maintenance treatment period - Tralokinumab Q4W (Experimental): Week 16 to Week 52:
  Tralokinumab responders from the initial treatment period re-randomised at Week 16 and administered tralokinumab maintenance subcutaneous injection regimen Q4W for 36 weeks.
  Subjects in this group receive alternating doses of tralokinumab SC injection and placebo SC injection every 2 weeks.
  Interventions: Drug: Tralokinumab; Drug: Placebo
- Maintenance treatment period - Placebo Q2W (Placebo Comparator): Week 16 to Week 52:
  Tralokinumab responders from initial treatment period randomised at Week 16 and administered placebo subcutaneous maintenance injection for 36 weeks.
  Interventions: Drug: Placebo
- Maintenance treatment period - Placebo (Placebo Comparator): Week 16 to Week 52:
  Placebo responders from the initial treatment period re-assigned at Week 16 and administered placebo maintenance subcutaneous injection regimen Q2W for 36 weeks.
  Interventions: Drug: Placebo
- Open-label treatment - Tralokinumab + optional TCS (Experimental): Week 16 to Week 52:
  Subjects receiving initial treatment with tralokinumab Q2W or placebo Q2W assigned to open-label treatment at Week 16 and administered Tralokinumab subcutaneous (SC) injection + optional TCS* regimen Q2W.
  OR
  Subjects receiving maintenance treatment with tralokinumab Q2W/Q4W or placebo assigned to open-label treatment after Week 16 and administered tralokinumab SC injection + optional TCS* regimen Q2W.
  *TCS = topical corticosteroids.
  Interventions: Drug: Tralokinumab
- Open-label short-term- Tralokinumab + optional TCS (Experimental): Week 52 to Week 68 [Short term extension (Japan only)] :
  Japanese subjects who were transferred to the open-label tralokinumab Q2W arm at Week 16 continued an additional 16 weeks (Week 52 to Week 66) of open-label treatment to receive 52 weeks of active therapy.
  Interventions: Drug: Tralokinumab

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous (SC) administration
  Arms: Initial treatment period - Tralokinumab Q2W; Maintenance treatment period - Tralokinumab Q2W; Maintenance treatment period - Tralokinumab Q4W; Open-label short-term- Tralokinumab + optional TCS; Open-label treatment - Tralokinumab + optional TCS
Drug: Placebo — Placebo contains the same excipients, in the same concentration only lacking tralokinumab
  Arms: Initial treatment period - Placebo Q2W; Maintenance treatment period - Placebo; Maintenance treatment period - Placebo Q2W; Maintenance treatment period - Tralokinumab Q4W

SUMMARY:
Primary objective:

To evaluate the efficacy of tralokinumab compared with placebo in treating moderate to severe atopic dermatitis (AD).

Secondary objectives:

To evaluate the efficacy of tralokinumab on severity and extent of AD, itch, and health related quality of life compared with placebo.

Maintenance objective:

To evaluate maintenance of effect with continued tralokinumab dosing up to 52 weeks compared to placebo for subjects achieving clinical response at Week 16.

DETAILED DESCRIPTION:
Subjects found eligible following the screening period were randomized 3:1 to initial treatment with tralokinumab 300 mg every 2 weeks (Q2W) or placebo. Randomization was stratified by region (North America, Europe, and Japan) and disease severity (Investigator's Global Assessment [IGA] 3 or 4).

Subjects achieving a clinical response at Week 16 (defined as IGA of 0 or 1 on a 5-point scale ranging from 0 [clear] to 4 [severe], or at least 75% reduction in Eczema Area and Severity Index [EASI] score from baseline [EASI75]) continued into maintenance treatment that continued until Week 52.

Subjects randomized to tralokinumab in the initial treatment period and who achieved a clinical response at Week 16 (defined by IGA 0 or 1, or EASI75) were re-randomized 2:2:1 to one of the following Q2W maintenance regimens stratified by region (North America, Europe, and Japan) and IGA response at Week 16 (IGA 0/1 or IGA >1):

* Tralokinumab 300 mg Q2W.
* Tralokinumab 300 mg Q4W (alternating dose administrations tralokinumab 300 mg and placebo).
* Placebo (Subjects randomized to placebo in the initial treatment period who achieved a clinical response at Week 16 [defined by IGA 0 or 1, or EASI75] continued to receive placebo Q2W in the maintenance treatment period).

Subjects not achieving a clinical response at Week 16 as well as those who met the criteria listed below during maintenance treatment were transferred to open-label tralokinumab 300 mg Q2W treatment with optional use of topical corticosteroid (TCS) up to Week 52.

Transfer to open-label treatment during maintenance:

Subjects with IGA=0 at Week 16: IGA of at least 2 and not achieved EASI75 over at least a 4-week period (i.e. over 3 consecutive visits).

Subjects with IGA=1 at Week 16: IGA of at least 3 and not achieved EASI75 over at least a 4-week period (i.e. over 3 consecutive visits).

Subjects with IGA >1 at Week 16: not achieved EASI75 over at least a 4-week period (i.e. over 3 consecutive visits).

Subjects transferring to open-label treatment had the option to self-administer tralokinumab in their home after adequate training (at 3 dosing visits in the open-label period after additional consent has been obtained) by site staff at the investigator's discretion.

After completion of the maintenance treatment period (or open-label treatment), all subjects, except for those who entered the open-label long-term extension trial, continued in a 14-week off-treatment follow-up period for the assessment of safety and anti-drug antibody (ADA).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorisation obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Age 18 and above.
3. Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD (34; Appendix 5).
4. Diagnosis of AD for ≥1 year.
5. Subjects who have a recent history (within 1 year before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable (e.g., due to important side effects or safety risks).

   Inadequate response is defined as failure to achieve and maintain remission or a low disease activity state (comparable to IGA 0=clear to 2=mild) despite treatment with a daily regimen of TCS of medium to higher potency (±TCI as appropriate), applied for at least 28 days or for the maximum duration recommended by the product prescribing information (e.g., 14 days for super potent TCS), whichever is shorter.

   Subjects with documented systemic treatment for AD in the past year are also considered as inadequate responders to topical treatments and are potentially eligible for treatment with tralokinumab after appropriate washout.

   Important side effects or safety risks are those that outweigh the potential treatment benefits and include intolerance to treatment, hypersensitivity reactions, significant skin atrophy, and systemic effects, as assessed by the investigator or by the subject's treating physician.
6. AD involvement of ≥10% body surface area at screening and baseline (visit 3).
7. An EASI score of ≥12 at screening and 16 at baseline.
8. An IGA score of ≥3 at screening and at baseline.
9. A Worst Daily Pruritus numeric rating scale (NRS) average score of ≥4 during the week prior to baseline.

   Worst Daily Pruritus NRS at baseline will be calculated from daily assessments of worst itch severity (Worst Daily Pruritus NRS) during the 7 days immediately preceding randomisation (Day 6 to 0). A minimum of 4 Worst Daily Pruritus NRS scores out of the 7 days is required to calculate the baseline average score. For subjects who do not have at least 4 scores reported during the 7 days immediately preceding the planned randomisation date, randomisation should be postponed until this requirement is met, but without exceeding the 6 weeks maximum duration for screening.
10. Subjects must have applied a stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation (refer to exclusion criterion no. 8 for limitations regarding emollients).
11. Women of childbearing potential must use a highly effective* form of birth control (confirmed by the investigator) throughout the trial and at least for 16 weeks (5 half lives) after last administration of IMP.

    * A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year) such as bilateral tubal occlusion, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), sexual abstinence (when this is in line with the preferred and usual life style of the subject), vasectomised partner (given that the subject is monogamous). The subjects must have used the contraceptive method continuously for at least 1 month prior to the pregnancy test at baseline. A female is defined as not being of child-bearing potential if she is postmenopausal (at least 12 months with no menses without an alternative medical cause prior to screening), or surgically sterile (hysterectomy, bilateral salpingectomy or bilateral oophorectomy).

Exclusion Criteria:

1. Concurrent enrolment in another clinical trial where the subject is receiving an IMP.
2. Previous randomisation in tralokinumab trials.
3. Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment, such as scabies, cutaneous lymphoma, or psoriasis.
4. Known active allergic or irritant contact dermatitis that is likely to interfere with the assessment of severity of AD.
5. Use of tanning beds or phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), within 6 weeks prior to randomisation.
6. Treatment with the following medications within 4 weeks prior to randomisation:

   * Systemic immunosuppressive/immunomodulating drugs (e.g. methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, Janus kinase inhibitors etc.).
   * Systemic corticosteroid use (excludes topical, inhaled, or intranasal delivery).
   * Three or more bleach baths during any week within the 4 weeks.
7. Treatment with the following medications within 2 weeks prior to randomisation

   * TCS.
   * TCI.
   * Topical PDE 4 inhibitor.
8. Initiation of treatment of AD with prescription emollients or emollients containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (subjects may continue using stable doses of such emollients if initiated before the screening visit).
9. Receipt of live attenuated vaccines 30 days prior to the date of randomisation and during the trial including the safety follow-up period.

   • Receipt of inactive/killed vaccinations (e.g. inactive influenza) are allowed, provided they are not administered within 5 days before/after any study visit.
10. Receipt of any marketed (i.e. immunoglobulin, anti-IgE) or investigational biologic agent, including dupilumab:

    * Any cell-depleting agents including but not limited to rituximab: within 6 months prior to randomisation, or until lymphocyte count returns to normal, whichever is longer.
    * Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to randomisation.
11. Receipt of any investigational non-biologic agent within 5 half-lives prior to randomisation.
12. Receipt of blood products within 4 weeks prior to screening.
13. Major surgery within 8 weeks prior to screening, or planned in-patient surgery or hospitalisation during the trial period.
14. Known or suspected allergy or reaction to any component of the IMP formulation.
15. History of any active skin infection within 1 week prior to randomisation.
16. History of a clinically significant infection within 4 weeks prior to randomisation which, in the opinion of the investigator or sponsor's medical expert, may compromise the safety of the subject in the trial, interfere with evaluation of the IMP, or reduce the subject's ability to participate in the trial. Clinically significant infections are defined as:

    * a systemic infection.
    * a serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
17. A helminth parasitic infection within 6 months prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy.
18. History of anaphylaxis following any biologic therapy.
19. History of immune complex disease.
20. History of cancer:

    * Subjects who have had basal cell carcinoma, localised squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
    * Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
21. Tuberculosis requiring treatment within the 12 months prior to screening. Evaluation will be according to local guidelines as per local standard of care.
22. History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the subject taking antiretroviral medications as determined by medical history and/or subject's verbal report.
23. History of chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance as judged by the investigator.
24. History of attempted suicide or is at significant risk of suicide (either in the opinion of the investigator or defined as a "yes" to suicidal ideation questions no. 4 or 5 or answering "yes" to suicidal behaviour on the Columbia-Suicide Severity Rating Scale [C-SSRS] Screening version).
25. Any disorder, including but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, immunological, psychiatric, or major physical impairment that is not stable, in the opinion of the investigator, and could:

    * Affect the safety of the subject throughout the trial.
    * Influence the findings of the trial or their interpretations.
    * Impede the subject's ability to complete the entire duration of trial.
26. Any clinically significant abnormal findings in physical examination, vital signs, electrocardiogram (ECG), haematology, clinical chemistry, or urinalysis during the screening period, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the trial, or may influence the results of the trial, or the subject's ability to complete entire duration of the trial.
27. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.0 times the ULN (upper limit of normal) at screening.
28. Positive hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb) or hepatitis C virus antibody (anti-HCV) serology at screening. Subjects with positive HBsAb may be randomised provided they are hepatitis B vaccinated and have negative HBsAg and HBcAb.
29. Subjects who are not willing to abstain from donating blood and/or plasma from the time of informed consent and for 16 weeks (5 half-lives) after last dose of IMP.
30. Subjects who are legally institutionalised.
31. Pregnant, breastfeeding, or lactating women.
32. Employees of the trial site or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wollenberg, Prof. Dr. med., Principal Investigator — Department of Dermatology and Allergy, Ludwig-Maximilian University Munich, Germany
Locations (123):
- United States (44):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Tien Q. Nguyen, MD, Inc., Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Quest Dermatology Research, Northridge, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - University Clinical Trials, Inc., San Diego, California
  - The GWU Medical Faculty Associates, Washington D.C., District of Columbia
  - Skin Care Research, Inc., Boca Raton, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - ACRC Dermatology, West Palm Beach, Florida
  - Georgia Pollens Clinical Research Centers, Inc., Albany, Georgia
  - Allergy Center at Brookstone Research, Columbus, Georgia
  - Dermatologic Surgery Specialists, Macon, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - PMG Research of Christie Clinic, Chicago, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - DermAssociates, PC, Rockville, Maryland
  - Clarkston Skin Research, Clarkston, Michigan
  - Derm Center, Troy, Michigan
  - MediSearch LLC, Saint Joseph, Missouri
  - JDR Dermatology Research, Las Vegas, Nevada
  - University at Buffalo Department of Dermatology, Buffalo, New York
  - Weil Cornell Medicine, New York, New York
  - Juva Skin & Laser Center, New York, New York
  - Deramatology Consulting Services, PLLC, High Point, North Carolina
  - Dermatologists of Greater Columbus, Bexley, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Health & Sciences University, Portland, Oregon
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Austin Dermatology Associates, Austin, Texas
  - Tekton Research, Austin, Texas
  - Dermtology Treatment and Research Center, Dallas, Texas
  - Houston Skin Associates, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
  - West Virginia Research Institute, Morgantown, West Virginia
- France (14):
  - Centre Hospitalier de Valence, Valence, Drôme
  - Hôpital St ANDRE, CHU de BORDEAUX, Service de Dermatologie, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Service de Dermatologie, Brest
  - CHU de Dijon, Service de Dermatologie, Dijon
  - Hôpital Claude Huriez-CHRU, Service de dermatologie, Lille
  - Hôpital Saint vincent de paul, Clinique de Dermatologie, Lille
  - Cabinet Médical, Le Bateau Blanc-Immeuble A, Martigues
  - GHRMSA, Service de Dermatologie, Mulhouse
  - Centre Hospitalier Universitaire, Clinique dermatologique 7 eme nord, Nantes
  - Hôpital de l'Archet II, Service de Dermatologie- Vénérologie, Nice
  - Hôpital Robert Debré, Service de Dermatologie, Reims
  - Hôpital Charles Nicolle, Clinique Dermatologique, Rouen
  - C.H.U. de Saint-Etienne - Hôpital Nord, Service de dermatologie, Saint-Etienne
  - CHU de Toulouse Hôpital Larrey, Service de Dermatologie, Toulouse
- Germany (22):
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen, Baden-Wurttemberg
  - Klinikum Augsburg, Klinik für Dermatologie und Allergologie, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen, Bavaria
  - LMU München, Klinik und Poliklinik für Dermatologie und Allergologie, München, Bavaria
  - Facharztpraxis für Dermatologie, Allergologie, Venerologie und Umweltmedizin, Mahlow, Brandenburg
  - Klinikum Darmstadt GmbH, Hautklinik, Darmstadt, Hessia
  - Hautärzte Zentrum Hannover, Hannover, Lower Saxony
  - Medizinische Hochschule Hannover, Klinik für Dermatologie, Allergologie und Venerologie, Hannover, Lower Saxony
  - KliFOs - Klinische Forschung Osnabrück, Osnabrück, Lower Saxony
  - Klinikum Bielefeld Rosenhöhe, Hautklinik, Bielefeld, North Rhine-Westphalia
  - Niesmann, Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Klinik und Poliklinik für Dermatologie und Allergologie, Bonn, North Rhine-Westphalia
  - Hautzentrum Dülmen, Dülmen, North Rhine-Westphalia
  - Universitätsklinikum Essen (AöR), Klinik für Dermatologie, Venerologie und Allergologie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster Klinik und Poliklinik für Hautkrankheiten Münster, Zentrale Studienkoordination für innovative Dermatologie, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Dermatologie, Dresden, Saxony
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Leipzig, Saxony
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Dermatologie und Venerologie, Halle, Saxony-Anhalt
  - SRH Wald-Klinikum Gera, Klinik für klinische Studien, Gera, Thuringia
  - Charité - Universitätsmedizin Berlin, Klinik für Dermatologie, Allergologie und Venerologie, Berlin
  - CMB Collegium Medicum Berlin GmbH, Berlin
  - SCIderm GmbH, Hamburg
- Japan (29):
  - Meiwa Hospital, Hyōgo, Nishinomiya
  - Hyogo College Of Medicine Hospital, Hyōgo, Nishinomiya
  - KUME Clinic, Sakai, Osaka
  - NTT Medical Center Tokyo, Tokyo, Shinagawa
  - Asahikawa City Hospital, Asahikawa
  - JR Sapporo Hospital, Chūō
  - Medical Corporation Kojinkai, Chūō
  - Fukuoka University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gifu University Hospital, Gifu
  - Osaka Habikono Medical Center, Habikino
  - Hamamatsu University hospital, Hamamatsu
  - Ichinomiya Municipal Hospital, Ichinomiya
  - Kagoshima University Hospital, Kagoshima
  - Kyoto Prefectural Hospital, Kyoto
  - Iwate Prefectural Central Hospital, Morioka
  - Chukyo Hospital, Nagoya
  - Takagi Dermatological Clinic, Obihiro
  - Gokeikai Osaka Kaisei Hospital, Ōsaka
  - Osaka Hospital, Ōsaka
  - Jichi Medical University Hospital, Tochigi
  - Tokyo Teishin Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - The Fraternity Memorial Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Ogikubo Hospital, Tokyo
  - Shirasaki Dermatology Clinic, Tōyama
- Spain (14):
  - Hospital Reina Sofía, Servicio Dermatología, Córdoba, Andalusia
  - Hospital Virgen de la Macarena, Servicio Dermatología, Seville, Andalusia
  - Hospital de Basurto, Servicio Dermatología, Bilbao, Basque Country
  - Hospital de Cruces, Servicio Dermatología, Bilbao, Basque Country
  - Hospital Germans Trias i Pujol, Servicio Dermatología, Badalona, Catalonia
  - Hospital Clinic de Barcelona, Dermatology Department, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Servicio Dermatología, Barcelona, Catalonia
  - Hospital del Mar, Servicio Dermatología, Barcelona, Catalonia
  - Clínica Universitaria de Navarra, Servicio Dermatología, Pamplona, Navarre
  - Hospital de Fuenlabrada, Servicio Dermatología, Madrid
  - Hospital Infanta Leonor, Servicio Dermatología, Madrid
  - Hospital Universitario de la Princesa, Servicio Dermatología, Madrid
  - Hospital Universitario La Paz, Servicio Dermatología, Madrid
  - Hospital Universitario y Politécnico La Fe, Servicio Dermatología, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayo T, Silverberg JI, Armstrong A, Guttman-Yassky E, Blauvelt A, Esdaile B, Kabashima K, Gooderham M, Kircik L, Schneider S, Bennike N, von Eyben R, Martel BC, Ropke MA, Katoh N, Alexis AF. Efficacy and Safety of Tralokinumab Across Racial Subgroups in Adults with Moderate-to-Severe Atopic Dermatitis: Post Hoc Analysis of Phase III Trials. Am J Clin Dermatol. 2025 Oct 21. doi: 10.1007/s40257-025-00985-1. Online ahead of print. PMID 41118053
- [Derived] Paller AS, Soong W, Boguniewicz M, Geng B, Thyssen JP, Bennike N, Schneider S, Wollenberg A. Effect of tralokinumab on moderate-to-severe atopic dermatitis in patients with atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Oct;135(4):425-433.e4. doi: 10.1016/j.anai.2025.06.022. Epub 2025 Jun 22. PMID 40555305
- [Derived] Chovatiya R, Ribero S, Wollenberg A, Park CO, Silvestre JF, Hong HC, Seneschal J, Saeki H, Thyssen JP, Oland CB, Gjerum L, Maslin D, Blauvelt A. Long-Term Disease Control and Minimal Disease Activity of Head and Neck Atopic Dermatitis in Patients Treated with Tralokinumab up to 4 Years. Am J Clin Dermatol. 2025 Jul;26(4):587-601. doi: 10.1007/s40257-025-00931-1. Epub 2025 Mar 14. PMID 40085349
- [Derived] Guttman-Yassky E, Kabashima K, Staumont-Salle D, Nahm WK, Pauser S, Da Rosa JC, Martel BC, Madsen DE, Ropke M, Arlert P, Steffensen L, Blauvelt A, Reich K. Targeting IL-13 with tralokinumab normalizes type 2 inflammation in atopic dermatitis both early and at 2 years. Allergy. 2024 Jun;79(6):1560-1572. doi: 10.1111/all.16108. Epub 2024 Apr 2. PMID 38563683
- [Derived] Simpson EL, Blauvelt A, Silverberg JI, Cork MJ, Katoh N, Mark T, Schneider SKR, Wollenberg A. Tralokinumab Provides Clinically Meaningful Responses at Week 16 in Adults with Moderate-to-Severe Atopic Dermatitis Who Do Not Achieve IGA 0/1. Am J Clin Dermatol. 2024 Jan;25(1):139-148. doi: 10.1007/s40257-023-00817-0. Epub 2023 Oct 7. PMID 37804473
- [Derived] Simpson EL, Pink AE, Blauvelt A, Gooderham M, Armstrong AW, Worm M, Katoh N, Peris K, Puig L, Barbarot S, Mark T, Steffensen LA, Tindberg AM, Wollenberg A. Tralokinumab Efficacy Over 1 Year in Adults with Moderate-to-Severe Atopic Dermatitis: Pooled Data from Two Phase III Trials. Am J Clin Dermatol. 2023 Nov;24(6):939-952. doi: 10.1007/s40257-023-00806-3. Epub 2023 Sep 8. PMID 37682422
- [Derived] Beck LA, Bieber T, Weidinger S, Tauber M, Saeki H, Irvine AD, Eichenfield LF, Werfel T, Arlert P, Jiang L, Ropke M, Paller AS. Tralokinumab treatment improves the skin microbiota by increasing the microbial diversity in adults with moderate-to-severe atopic dermatitis: Analysis of microbial diversity in ECZTRA 1, a randomized controlled trial. J Am Acad Dermatol. 2023 Apr;88(4):816-823. doi: 10.1016/j.jaad.2022.11.047. Epub 2022 Dec 5. PMID 36473633
- [Derived] Blauvelt A, Gooderham M, Bhatia N, Langley RG, Schneider S, Zoidis J, Kurbasic A, Armstrong A, Silverberg JI. Tralokinumab Efficacy and Safety, with or without Topical Corticosteroids, in North American Adults with Moderate-to-Severe Atopic Dermatitis: A Subanalysis of Phase 3 Trials ECZTRA 1, 2, and 3. Dermatol Ther (Heidelb). 2022 Nov;12(11):2499-2516. doi: 10.1007/s13555-022-00805-y. Epub 2022 Sep 24. PMID 36152216
- [Derived] Wollenberg A, Blauvelt A, Guttman-Yassky E, Worm M, Lynde C, Lacour JP, Spelman L, Katoh N, Saeki H, Poulin Y, Lesiak A, Kircik L, Cho SH, Herranz P, Cork MJ, Peris K, Steffensen LA, Bang B, Kuznetsova A, Jensen TN, Osterdal ML, Simpson EL; ECZTRA 1 and ECZTRA 2 study investigators. Tralokinumab for moderate-to-severe atopic dermatitis: results from two 52-week, randomized, double-blind, multicentre, placebo-controlled phase III trials (ECZTRA 1 and ECZTRA 2). Br J Dermatol. 2021 Mar;184(3):437-449. doi: 10.1111/bjd.19574. Epub 2020 Dec 30. PMID 33000465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening period was 2 to 6 weeks and included 1 or 2 visits. The exact duration depended on the wash-out period defined by the exclusion criteria. If no wash-out or only a 2-week wash-out was required, screening Visits 1 and 2 were combined. Eligibility was assessed at the (first) screening visit and on Day 0 prior to randomisation.
Groups:
- Initial Treatment Period - Tralokinumab 300 mg Q2W: Week 0 to Week 16:
  Tralokinumab 300 mg Q2W
  Tralokinumab: Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for SC administration
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Initial Treatment Period - Placebo Q2W: Week 0 to Week 16:
  Placebo Q2W
  Placebo: Placebo contains the same excipients, in the same concentration, only lacking tralokinumab.
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of placebo to receive a total loading dose (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of placebo.
- Maintenance Treatment Period - Tralokinumab 300 mg Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomised to tralokinumab re-randomised to tralokinumab 300 mg Q2W maintenance dosing regimen.
  At each visit, subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg tralokinumab.
- Maintenance Treatment Period - Tralokinumab 300 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomised to tralokinumab re-randomised to tralokinumab 300 mg Q4W maintenance dosing regimen.
  At each visit, subject received alternating dose administrations: 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab and 2 SC injections (each 1.0 mL) of placebo.
- Maintenance Treatment Period - Placebo Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomised to tralokinumab re-randomised to placebo Q2W dosing regimen.
  At each visit, each subject received 2 SC injections (each 1.0 mL) of placebo Q2W to receive a total dose of placebo.
- Maintenance Treatment Period- Placebo Q2W - Tralokinumab Naive: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomized to placebo re-assigned to placebo Q2W.
  At each visit, subject received 2 SC injections (each 1.0 mL) of placebo Q2W to receive a total dose of placebo.
- Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS: Week 16 to Week 52:
  Subjects receiving initial treatment with tralokinumab/placebo Q2W who did not achieve protocol-defined clinical response assigned to open-label treatment at Week 16 with tralokinumab 300 mg Q2W regimen + optional topical corticosteroids (TCS) OR Subjects receiving maintenance treatment with tralokinumab 300 mg Q2W/Q4W or placebo Q2W assigned to open-label treatment after Week 16 with tralokinumab 300 mg Q2W regimen + optional TCS if
  * IGA of at least 2 and not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA=0 at Week 16 OR
  * IGA of at least 3 and not achieving EASI75 over at least a 4-week period (i.e. over 3 consecutive visits) for subjects with IGA=1 at Week 16 OR
  * Not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA>1 at Week 16
  At each visit, subjects received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg.
- Open-label Treatment - Tralokinumab 300 mg Q2W + Optional TCS: Week 52 to Week 66 [Short term extension (Japan only)]:
  Japanese subjects who did not achieve protocol-defined clinical response assigned to open-label treatment at Week 16 with tralokinumab 300 mg Q2W regimen + optional topical corticosteroids (TCS) continued an additional 16 weeks (Week 52 to Week 66) of open-label treatment to receive 52 weeks of active therapy.
  At each visit, subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg.
Period: Initial Treatment Period
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Placebo Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Maintenance Treatment Period- Placebo Q2W - Tralokinumab Naive | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS | Open-label Treatment - Tralokinumab 300 mg Q2W + Optional TCS
Started | 603 | 199 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 550 | 179 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 53 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not dosed | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued IMP before Week 16 | 51 | 18 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label Treatment
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Placebo Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Maintenance Treatment Period- Placebo Q2W - Tralokinumab Naive | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS | Open-label Treatment - Tralokinumab 300 mg Q2W + Optional TCS
Started (Open-label treatment period was in parallel to the maintenance treatment period.) | 0 | 0 | 0 | 0 | 0 | 0 | 564 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 446 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 118 | 0
Not completed — Discontinued IMP | 0 | 0 | 0 | 0 | 0 | 0 | 112 | 0
Not completed — Completed Week 50 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Period: Maintenance Treatment Period
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Placebo Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Maintenance Treatment Period- Placebo Q2W - Tralokinumab Naive | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS | Open-label Treatment - Tralokinumab 300 mg Q2W + Optional TCS
Started (Maintenance treatment period was in parallel to the open-label treatment period.) | 0 | 0 | 71 | 78 | 36 | 29 | 0 | 0
Completed | 0 | 0 | 44 | 53 | 21 | 15 | 0 | 0
Not Completed | 0 | 0 | 27 | 25 | 15 | 14 | 0 | 0
Not completed — Not dosed | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Discontinued IMP | 0 | 0 | 3 | 5 | 4 | 4 | 0 | 0
Not completed — Transfer to open-label treatment | 0 | 0 | 21 | 18 | 9 | 10 | 0 | 0
Not completed — Completed Week 50 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Open-label (Short Term Extension)
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Placebo Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Maintenance Treatment Period- Placebo Q2W - Tralokinumab Naive | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS | Open-label Treatment - Tralokinumab 300 mg Q2W + Optional TCS
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 65
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Discontinued IMP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Initial Treatment Period - Tralokinumab 300 mg Q2W: Week 0 to Week 16:
  Tralokinumab 300 mg Q2W
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Initial Treatment Period - Placebo Q2W: Week 0 to Week 16:
  Placebo Q2W
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of placebo to receive a total loading dose (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of placebo.
- Total: Total of all reporting groups
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Placebo Q2W | Total
Number analyzed (Participants) | 603 | 199 | 802
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.7) | 39.4 (15.2) | 38.8 (14.1)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 574 | 185 | 759
  65-84 years | 28 | 14 | 42
  >=85 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 76 | 328
  Male | 351 | 123 | 474
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 17 | 70
  Not Hispanic or Latino | 548 | 179 | 727
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 426 | 138 | 564
  Black or african american | 41 | 18 | 59
  Asian | 120 | 40 | 160
  American indian or alaska native | 1 | 0 | 1
  Native hawaiian or other pacific islander | 5 | 0 | 5
  Other | 8 | 0 | 8
  Missing | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 149 | 49 | 198
  Japan | 96 | 31 | 127
  France | 85 | 23 | 108
  Germany | 200 | 73 | 273
  Spain | 73 | 23 | 96
Investigator's Global Assessment [Count of Participants; unit: Participants] — The Investigator's Global Assessment (IGA) is an instrument used in clinical trials to rate the severity of the subject's global atopic dermatitis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 296 | 95 | 391
    Severe | 305 | 102 | 407
    Missing | 2 | 2 | 4
Eczema Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Eczema Area and Severity Index (EASI) is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition. Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 601 | 197 | 798
    (all) | 32.2 (13.7) | 32.9 (13.9) | 32.4 (13.8)
Scoring Atopic Dermatitis [Mean (Standard Deviation); unit: units on a scale] — The Scoring Atopic Dermatitis (SCORAD) is a validated tool to evaluate the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with higher values indicating more extensive and/or severe condition. Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 601 | 197 | 798
    (all) | 70.3 (13.0) | 71.7 (12.5) | 70.6 (12.9)
Dermatology Life Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Dermatology Life Quality Index (DLQI) consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their health-related quality of life (HQoL) over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all ⁄not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor HQoL. Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 591 | 194 | 785
    (all) | 16.8 (7.1) | 17.0 (6.6) | 16.9 (7.0)
Worst Daily Pruritus NRS (weekly average) [Mean (Standard Deviation); unit: units on a scale] — Subjects assess their worst itch severity over the past 24 hours using an 11-point NRS ('Worst Daily Pruritus NRS') with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'. Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 598 | 195 | 793
    (all) | 7.7 (1.4) | 7.7 (1.4) | 7.7 (1.4)
Body surface area affected by atopic dermatitis (AD) [Mean (Standard Deviation); unit: percentage affected] — Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  percentage affected
    number analyzed (Participants) | 603 | 198 | 801
    (all) | 52.7 (24.1) | 54.2 (25.6) | 53.1 (24.5)
Age of onset of atopic dermatitis (AD) [Median (Inter-Quartile Range); unit: years] — Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  years
    number analyzed (Participants) | 603 | 198 | 801
    (all) | 3.0 [1.0 to 14.0] | 3.0 [0.0 to 13.0] | 3.0 [0.0 to 13.0]
Duration of atopic dermatitis (AD) [Mean (Standard Deviation); unit: years] — Population: Number of subjects analysed = subjects with available data for the baseline parameter.
  years
    number analyzed (Participants) | 603 | 198 | 801
    (all) | 27.9 (14.5) | 29.6 (15.1) | 28.3 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: At Week 16
Population: The full analysis set (FAS: all subjects randomised to initial treatment who were exposed to IMP) was used for the primary analysis; 802 subjects were randomised to initial treatment and 798 received IMP, thus the FAS comprised of 798 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab 300 mg Q2W: Week 0 to Week 16:
  Tralokinumab 300 mg Q2W
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Placebo Q2W: Week 0 to Week 16:
  Placebo Q2W
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of placebo to receive a total loading dose (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of placebo.
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 95 | 14
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity.The null hypothesis of no difference in response rates between tralokinumab and placebo were tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoints tested sequentially at a 5% significance level; p = 0.002, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'. Subjects with missing data or subjects who received rescue medication prior to Week 16 were considered non-responders; Primary endpoints tested sequentially at a 5% significance level; Risk Difference (RD) = 8.6, 95% CI 2-sided [4.1 to 13.1] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

2. Primary Outcome: Subjects Achieving at Least 75% Reduction in Eczema Area and Severity Index [EASI] at Week 16
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Time Frame: At Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 150 | 25
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rates between tralokinumab and placebo were tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoints tested sequentially at a 5% significance level; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Primary endpoints tested sequentially at a 5% significance level; Risk Difference (RD) = 12.1, 95% CI 2-sided [6.5 to 17.7] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

3. Secondary Outcome: Reduction of Worst Daily Pruritus Numeric Rating Scale (Weekly Average) of at Least 4 From Baseline to Week 16.
Description: Subjects will assess their worst itch severity over the past 24 hours using an 11 point NRS ('Worst Daily Pruritus NRS') with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
Time Frame: Week 0 to Week 16
Population: Full analysis set (FAS). Number of subjects analysed = subjects with baseline pruritus NRS weekly average ≥4.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 594 | 194
Participants | 119 | 20
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Reduction of Worst Daily Pruritus NRS weekly average ≥4 at Week 16 was tested after the sequential testing of IGA 0/1 and EASI75 if these tests showed statistical significance; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'Composite', subjects who received rescue medication prior to Week 16 or have missing data at Week 16 were considered as non-responders; Tested sequentially at a 5% significance level; Risk Difference (RD) = 9.7, 95% CI 2-sided [4.4 to 15] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

4. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with higher values indicating a more extensive and/or severe condition.
Time Frame: Week 0 to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
units on a scale | -25.2 (0.94) | -14.7 (1.80)
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Data collected after permanent discontinuation of IMP or after initiation of rescue medication were not included in the analysis; Test type: Superiority — Multiplicity adjustment using the Holm method; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'. Repeated measurements model on post-baseline data. In case of no post-baseline assessments before initiation of rescue medication, the Week 2 change was imputed as 0; Difference of least square means = -10.4, 95% CI 2-sided [-14.4 to -6.5]

5. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Baseline to Week 16
Description: The Dermatology Life Quality Index (DLQI) is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their quality of life (QoL) over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4 point Likert scale (0 = not at all ⁄not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor QoL.
Time Frame: Week 0 to Week 16
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
units on a scale | -7.1 (0.31) | -5.0 (0.59)
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Data collected after permanent discontinuation of IMP or initiation of rescue medication not included; Test type: Superiority — Multiplicity adjustment using Holm method; p = 0.002, Repeated measurements model — [p-value comment as in outcome 4, analysis 1]; Difference of least square means = -2.1, 95% CI 2-sided [-3.4 to -0.8]

6. Secondary Outcome: Subjects With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 52 Among Subjects With IGA of 0/1 at Week 16
Description: as for outcome 1
Time Frame: At Week 52
Population: Maintenance analysis set - Subjects who achieved IGA 0/1 at Week 16 after initial treatment with tralokinumab without use of rescue medication.
  Subjects who were treated with placebo during initial treatment period (tralokinumab naïve arm) and who continued to the maintenance period were not part of the analysis of maintenance endpoints and therefore this arm is not included for outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab 300 mg Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to tralokinumab 300 mg Q2W maintenance dosing regimen.
  At each visit, subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg tralokinumab.
- Tralokinumab 300 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to tralokinumab 300 mg Q4W maintenance dosing regimen.
  At each visit, subject received alternating dose administrations: 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab and 2 SC injections (each 1.0 mL) of placebo.
- Placebo Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to placebo Q2W dosing regimen.
  At each visit, subject received 2 SC injections (each 1.0 mL) of placebo Q2W to receive a total dose of placebo.
Arm/Group | Tralokinumab 300 mg Q2W | Tralokinumab 300 mg Q4W | Placebo Q2W
Number analyzed (Participants) | 39 | 36 | 19
Participants | 20 | 14 | 9
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Testing according to the hierarchical testing procedure in the order: IGA 0/1 at Week 52 between Q2W vs Placebo, EASI75 at Week 52 between Q2W vs Placebo, IGA 0/1 at Week 52 between Q4W vs Placebo, and EASI75 at Week 52 between Q4W vs Placebo; Test type: Superiority; p = 0.68, Cochran-Mantel-Haenszel — Based on the primary analysis of the 'composite' estimand. Subjects who received rescue medication or were transferred to open-label treatment were considered non-responders. P value was considered non-significant; This test was not statistically significant and hence next maintenance endpoint in the sequential testing procedure was not evaluated; Risk Difference (RD) = 6.0, 95% CI 2-sided [-21.8 to 33.7] — Mantel-Haenszel risk difference compared to placebo, stratified by region
Statistical Analysis 2: Comparison: Tralokinumab 300 mg Q4W vs Placebo Q2W; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.50, Cochran-Mantel-Haenszel — Test not evaluated for significance. Based on the primary analysis of the 'composite' estimand. Subjects who received rescue medication or were transferred to open-label treatment were considered non-responders; Risk Difference (RD) = -9.5, 95% CI 2-sided [-37.1 to 18.0] — Mantel-Haenszel risk difference compared to placebo, stratified by region

7. Secondary Outcome: Subjects With at Least 75% Reduction in Eczema Area and Severity Index [EASI] at Week 52 Among Subjects With EASI75 at Week 16
Description: as for outcome 2
Time Frame: At Week 52
Population: Maintenance analysis set: Subjects who achieved EASI75 at Week 16 after inital treatment with tralokinumab without use of rescue medication.
  Subjects who were treated with placebo during initial treatment period (tralokinumab naïve arm) and who continued to the maintenance period were not part of the analysis of maintenance endpoints and therefore this arm is not included for outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab 300 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomised to tralokinumab 300 mg Q4W maintenance dosing regimen.
  At each visit, subject received alternating dose administrations: 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab and 2 SC injections (each 1.0 mL) of placebo.
Arm/Group | Tralokinumab 300 mg Q2W | Tralokinumab 300 mg Q4W | Placebo Q2W
Number analyzed (Participants) | 47 | 57 | 30
Participants | 28 | 28 | 10
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.056, Cochran-Mantel-Haenszel — Test not evaluated for significance. Based on the primary analysis of the primary estimand 'composite'. Subjects who received rescue medication or were transferred to open-label treatment are considered non-responders; Risk Difference (RD) = 21.2, 95% CI 2-sided [-0.2 to 42.6] — Mantel-Haenszel risk difference compared to placebo, stratified by region
Statistical Analysis 2: Comparison: Tralokinumab 300 mg Q4W vs Placebo Q2W; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.27, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 2]; Risk Difference (RD) = 11.7, 95% CI 2-sided [-8.7 to 32.0] — Mantel-Haenszel risk difference compared to placebo, stratified by region

8. Secondary Outcome: Safety and Tolerability: Adverse Event (AE) /Serious Adverse Event (SAE) Frequency
Description: Overall summary of AEs and SAEs during the Initial treatment period is presented. For list of AEs and SAEs by MedDRA system organ class (SOC) and preferred term (PT) during the entire trial period (including safety follow-up), see Adverse Events Overview section.
Time Frame: Week 0 to Week 16
Population: The analysis was performed on the safety analysis set. The safety analysis set comprised of participants who received at least 1 dose of IMP during the trial.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Q2W: Week 0 to Week 16:
  Placebo Q2W.
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of placebo to receive a total loading dose (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of placebo.
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 602 | 196
Participants
  AEs | 411 | 133
  SAEs | 23 | 8

9. Secondary Outcome: Frequency of Anti-drug Antibodies
Description: Anti-tralokinumab antibody levels were analysed using a validated bioanalytical method.
Time Frame: Week 0 to Week 16
Population: All subjects in the safety analysis set are included
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 602 | 196
Participants
  Total positive | 10 | 3
  Pre-existing | 0 | 2
  Treatment-boosted | 0 | 0
  Treatment emergent | 10 | 1
  Perishing | 5 | 3
  Negative | 564 | 177
  No post-baseline anti-drug antibody assessment | 23 | 13

10. Secondary Outcome: Subjects Achieving at Least 50% Reduction in Eczema Area and Severity Index [EASI] at Week 16
Description: as for outcome 2
Time Frame: At Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 250 | 42
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority — Based on the primary analysis of the primary estimand 'composite'. Subjects with missing data or subjects who received rescue medication prior to Week 16 were considered non-responders. The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.1, 95% CI 2-sided [13.3 to 26.8] — Mantel-Haenszel risk difference, stratified by region and disease severity

11. Secondary Outcome: Subjects Achieving at Least 90% Reduction in Eczema Area and Severity Index [EASI] at Week 16
Description: as for outcome 2
Time Frame: At Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 87 | 8
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'. Subjects with missing data or subjects who received rescue medication prior to Week 16 were considered non-responders. The statistical test was not controlled for multiplicity; Risk Difference (RD) = 10.3, 95% CI 2-sided [6.4 to 14.1] — Mantel-Haenszel risk difference, stratified by region and disease severity

12. Secondary Outcome: Change From Baseline to Week 16 in Eczema Area and Severity Index [EASI] Score
Description: as for outcome 2
Time Frame: Week 0 to Week 16
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
units on a scale | -15.5 [-16.6 to -14.4] | -9.0 [-11.1 to -7.0]
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Data collected after permanent discontinuation of IMP or initiation of rescue medication not included. In case of no post-baseline assessments before initiation of rescue medication, the Week 2 change will be imputed as 0; Test type: Superiority; p < 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference of least square means = -6.4, 95% CI 2-sided [-8.8 to -4.1]

13. Secondary Outcome: Subjects Achieving at Least 75% Reduction in Scoring Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with a higher values indicating a more extensive and/or severe condition.
Time Frame: At Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 53 | 6
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel — Based on the primary analysis of the 'composite' estimand. Subjects who received rescue medication prior to Week 16 or with missing data at Week 16 were considered nonresponders. The statistical test was not controlled for multiplicity; Risk Difference (RD) = 5.7, 95% CI 2-sided [2.5 to 8.9] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

14. Secondary Outcome: Subjects Achieving at Least 50% Reduction in Scoring Atopic Dermatitis (SCORAD) at Week 16
Description: as for outcome 4
Time Frame: At Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 601 | 197
Participants | 156 | 23
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the 'composite' estimand. Subjects who received rescue medication prior to Week 16 or with missing data at Week 16 were considered non-responders. The statistical test was not controlled for multiplicity; Risk Difference (RD) = 14.1, 95% CI 2-sided [8.6 to 19.6] — Mantel-Haenszel risk difference stratified by region and disease severity

15. Secondary Outcome: Change From Baseline to Week 16 in Worst Daily Pruritus NRS (Weekly Average)
Description: as for outcome 3
Time Frame: Week 0 to Week 16
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 598 | 195
units on a scale | -2.6 [-2.8 to -2.4] | -1.7 [-2.1 to -1.3]
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Data collected after permanent discontinuation of IMP or initiation of rescue medication not included. In case of no post-baseline assessments before initiation of rescue medication, the Week 1 change will be imputed as 0; Test type: Superiority; p < 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference of least square means = -0.9, 95% CI 2-sided [-1.4 to -0.4]

16. Secondary Outcome: Reduction of Worst Daily Pruritus NRS (Weekly Average) ≥3 From Baseline to Week 16
Description: as for outcome 3
Time Frame: Week 0 to Week 16
Population: Full analysis set. Number of subjects analysed = subjects with baseline Pruritus NRS weekly average of at least 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 597 | 195
Participants | 177 | 28
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Subjects who received rescue medication prior to Week 16 or have missing data at Week 16 were considered as non-responders. The statistical test was not controlled for multiplicity; Risk Difference (RD) = 15.2, 95% CI 2-sided [9.2 to 21.3] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

17. Secondary Outcome: Reduction From Baseline to Week 16 of Dermatology Life Quality Index (DLQI) of ≥4 Points Among Subjects With Baseline DLQI ≥4
Description: The DLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their QoL over the last week such as dermatology related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4 point Likert scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor QoL.
Time Frame: Week 0 to Week 16
Population: Full analysis set. Number of subjects analysed = subjects with baseline DLQI ≥4.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 578 | 190
Participants | 258 | 60
Statistical Analysis 1: Comparison: Tralokinumab 300 mg Q2W vs Placebo Q2W; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Risk Difference (RD) = 13.0, 95% CI 2-sided [5.4 to 20.5] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

ADVERSE EVENTS:
Time Frame: Initial Treatment Period: Week 0 to Week 16, Maintenance Treatment Period: Week 16 to Week 52, Open-label Treatment: Week 16 to Week 52; Safety Follow-up Period: Week 52 to Week 66 and Week 68 to Week 82 (for selected Japanese subjects).
Groups:
- Initial Period - Tralokinumab Q2W: Initial Period - Tralokinumab Q2W
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Initial Period - Placebo: Initial Period - Placebo
  At Day 0, each subject received 4 SC injections (each 1.0 mL) of placebo to receive a total loading dose (4.0 mL). At subsequent visits (Q2W) each subject received 2 SC injections (each 1.0 mL) of placebo.
- Maintenance Period - Tralokinumab Q2W: Maintenance Period - Tralokinumab Q2W
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to tralokinumab 300 mg Q2W maintenance dosing regimen.
  At each visit, subject received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg tralokinumab.
- Maintenance Period - Tralokinumab Q4W: Maintenance Period - Tralokinumab Q4W
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to tralokinumab 300 mg Q4W maintenance dosing regimen.
  At each visit, subject received alternating dose administrations: 2 SC injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab and 2 SC injections (each 1.0 mL) of placebo.
- Maintenance Period - Placebo: Maintenance Period - Placebo
  Subjects achieving a clinical response at Week 16 and initially randomized to tralokinumab re-randomized to placebo Q2W dosing regimen.
  At each visit, subject received 2 SC injections (each 1.0 mL) of placebo Q2W to receive a total dose of placebo.
- Maintenance Period - Placebo - Tralokinumab Naive: Maintenance Period - Placebo - Tralokinumab Naive
  Subjects achieving a clinical response at Week 16 and initially randomized to placebo re-assigned to placebo Q2W.
  At each visit, subject received 2 SC injections (each 1.0 mL) of placebo Q2W to receive a total dose of placebo.
- Open-label Period - Tralokinumab Q2W + Optional TCS: Open-label Period - Tralokinumab Q2W + Optional TCS
  Subjects receiving initial treatment with tralokinumab/placebo Q2W who did not achieve protocol-defined clinical response assigned to open-label treatment at Week 16 with tralokinumab 300 mg Q2W regimen + optional topical corticosteroids (TCS) OR Subjects receiving maintenance treatment with tralokinumab 300 mg Q2W/Q4W or placebo Q2W assigned to open-label treatment after Week 16 with tralokinumab 300 mg Q2W regimen + optional TCS if IGA of at least 2 and not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA=0 at Week 16 OR IGA of at least 3 and not achieving EASI75 over at least a 4-week period (i.e. over 3 consecutive visits) for subjects with IGA=1 at Week 16 OR Not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA>1 at Week 16 At each visit, subjects received 2 SC injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg.
- Safety Follow-up: Subjects who spent any amount of time in the safety follow-up period, independently of the treatment(s) received before. No treatment was administered to the subjects during the safety follow-up period. Eligible participants who completed treatment could transfer to an open-label long-term extension trial (conducted under a separate protocol) at any any time during the safety follow-up period.
Arm/Group | Initial Period - Tralokinumab Q2W | Initial Period - Placebo | Maintenance Period - Tralokinumab Q2W | Maintenance Period - Tralokinumab Q4W | Maintenance Period - Placebo | Maintenance Period - Placebo - Tralokinumab Naive | Open-label Period - Tralokinumab Q2W + Optional TCS | Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/602 | 0/196 | 0/68 | 0/76 | 0/35 | 0/29 | 0/563 | 0/595
Serious Adverse Events (participants affected / at risk) | 23/602 | 8/196 | 1/68 | 3/76 | 0/35 | 1/29 | 27/563 | 16/595
Other Adverse Events (participants affected / at risk) | 351/602 | 114/196 | 37/68 | 39/76 | 20/35 | 9/29 | 304/563 | 29/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Period - Tralokinumab Q2W (N=602) | Initial Period - Placebo (N=196) | Maintenance Period - Tralokinumab Q2W (N=68) | Maintenance Period - Tralokinumab Q4W (N=76) | Maintenance Period - Placebo (N=35) | Maintenance Period - Placebo - Tralokinumab Naive (N=29) | Open-label Period - Tralokinumab Q2W + Optional TCS (N=563) | Safety Follow-up (N=595)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accessory cardiac pathway (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leishmaniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Period - Tralokinumab Q2W (N=602) | Initial Period - Placebo (N=196) | Maintenance Period - Tralokinumab Q2W (N=68) | Maintenance Period - Tralokinumab Q4W (N=76) | Maintenance Period - Placebo (N=35) | Maintenance Period - Placebo - Tralokinumab Naive (N=29) | Open-label Period - Tralokinumab Q2W + Optional TCS (N=563) | Safety Follow-up (N=595)
Conjunctivitis allergic (Eye disorders) | 16 (16) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 13 (14) | 2 (2)
Injection site reaction (General disorders) | 24 (47) | 0 (0) | 5 (13) | 7 (21) | 1 (1) | 0 (0) | 28 (60) | 0 (0)
Bronchitis (Infections and infestations) | 11 (12) | 4 (4) | 3 (3) | 7 (8) | 2 (2) | 1 (1) | 14 (15) | 1 (1)
Conjunctivitis (Infections and infestations) | 43 (50) | 4 (4) | 3 (3) | 4 (6) | 0 (0) | 0 (0) | 41 (52) | 4 (4)
Influenza (Infections and infestations) | 18 (18) | 5 (5) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 7 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 15 (16) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 139 (172) | 41 (54) | 14 (17) | 18 (26) | 4 (5) | 2 (4) | 143 (201) | 12 (12)
Wrong patient received medication (Injury, poisoning and procedural complications) | 8 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Liver function test increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 18 (19) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 28 (50) | 10 (16) | 6 (12) | 2 (2) | 3 (6) | 0 (0) | 22 (29) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 10 (10) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 152 (198) | 75 (123) | 11 (14) | 14 (22) | 13 (18) | 6 (10) | 123 (201) | 10 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (41) | 10 (15) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 20 (27) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 18 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-centre publication within 18 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (2):
  • Study Protocol (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03131648/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03131648/SAP_001.pdf